

NCT05048433

Version Date: 07/31/2023

Study Contact: Timothy Walker, PhD Telephone:





# PARENTAL PERMISSION FOR CHILD PARTICIPATION SURVEY AND ACCELEROMETERS

**Study Title:** Developing and testing an implementation strategy for active learning to

promote physical activity in children

**Study Sponsor:** National Heart, Lung, and Blood Institute (NHLBI)

Principal Investigator: Timothy J. Walker, PhD, Assistant Professor

Study Contact: Office Phone – ; Email –

We are doing this research study to develop and test an implementation strategy to support the use of active learning approaches in elementary schools to increase students' physical activity levels. If you choose to allow your child to take part in this study, your child will be asked to complete a survey about their physical activity and opinions about doing physical movements as part of their classroom learning.

There is a possible risk of breach of confidentiality. There may be no direct benefit for you child being in the study; however, your taking part may help improve how physical activity can be supported in schools leading to better health and academic performance for youth.

Participation in this research study is voluntary. You may choose not to allow your child to take part in this research study or may choose to leave the research study at any time. Your decision will not change your child's status with their school.

If you are interested in participating, please continue reading below.

#### What is the purpose of this research study?

The study purpose is to test an implementation strategy to support the use of physically active learning in elementary schools to increase students' physical activity levels.

The National Heart, Lung, and Blood Institute (NHLBI) is paying UTHealth for their work on this study.

A description of this clinical trial will be available on <a href="http://www.clinicaltrials.gov">http://www.clinicaltrials.gov</a>, as required by U.S. Law. This will not include information that can identify your child. After the study has ended, website will include a summary of the results. You can search this website at any time.

### Who is being asked to take part in this study?

You are being asked to allow your child to take part in this research study because your child attends a school that is participating in the study. About 1,100 students from two different schools in Houston will take part in the study.

### What will happen if your child takes part in this study?

As part of the study, your child will be asked to complete questions about their physical activity and their opinions about being active during classroom time. These questions will be completed three times:

Study Contact: Timothy Walker, PhD

Telephone:

#UTHealth Houston IRB NUMBER: HSC-SPH-20-0861 IRB APPROVAL DATE: 07/31/2023

once at the start of the study, and 6 and 12 months from the start of the study. The school will also share your child's demographic, academic, fitness, and behavior data.

If you allow your child to take part in this study your child may be randomly selected to wear an accelerometer during school hours. There is a 20% chance your child will be selected to wear an accelerometer. An accelerometer is a device worn on a belt over the clothing that tracks movements to show how physically active your child is during the school day. The accelerometer is about the size of a large wrist watch (see example image). The accelerometer will be put on once your child arrives at school and removed the school and school and removed the school and scho



image). The accelerometer will be put on once your child arrives at school and removed prior to dismissal. The accelerometer will provide activity counts throughout the school day, which will be used to measure time spent being physically active during the school day.

## How long will your child be in the study?

The study will last about 1 year in total. If your child takes part in the study, his or her participation will last for 1 year and will involve completing a survey three times throughout the year (at the start of the study, and 6 and 12 months from the start of the study). In addition, your child may wear an accelerometer for 1-week during school hours three times throughout the year.

## What choices does your child have, other than this study?

There are no other options for your child if they choose not to participate in this study.

## What are the risks of taking part in this study?

There are minimal risks for study participation. There is a possible risk of breach of confidentiality. Or your child may not be comfortable wearing an activity tracking belt. You child can remove the belt at any time and does not have to answer any questions they are not comfortable answering.

### What are the benefits to taking part in this study?

There may be no direct benefit for you child being in the study. However, your child's participation may help improve how physical activity can be supported in schools leading to better health and academic performance for youth.

### Can your child stop taking part in this study?

You may decide to stop your child from taking part in the study at any time. To withdraw from the study, please contact Timothy Walker, PhD at If your child stops participating in this study, the information already collected will still be used in the data analysis. However, no further information will be collected without your permission.

While taking part in this study, the study team will notify you of new information that may become available and could affect your willingness to allow your child to stay in the study.

## What happens if your child is injured during the study?

If your child suffers an injury as a result of taking part in this research study, please understand that nothing has been arranged to provide free treatment of the injury or any other type of payment. However, necessary facilities, emergency treatment, and professional services will be available to your child, just as they are to the general community. You should report any such injury to Timothy Walker, PhD at You will not give up any of your child's legal rights by signing this consent form.

What are the costs of taking part in this study?

**Study Contact:** Timothy Walker, PhD

Telephone:



IRB NUMBER: HSC-SPH-20-0861 IRB APPROVAL DATE: 07/31/2023 There are not costs to participating in this study.

## How will your child's privacy and confidentiality be protected?

Your child's privacy is important and your child's participation in this study will be kept confidential. However, absolute confidentiality cannot be guaranteed.

Personal identifiers such as your child's name will be removed from the information and data records collected in this study. After we remove all identifiers, the information or data may be used for future research or shared with other researchers without your additional permission.

Please note that you do not have to sign this Authorization, but if you do not, your child may not participate in this research study.

| participate in this research | study. | | |
|---|---|---|---|
| Authorization, researchers necessary to maintain the in you must contact Timothy N | and revoke (take back) this And may still use information they integrity or reliability of the cullwalker in writing at the end of the color of the | already have obtained al rrent research. To revoke | bout your child as |
| If you have questions at any<br>, as he will be | ou have questions about the y time about this research stude glad to answer your question oice concerns, obtain informa | dy, please feel free to cor<br>is. You can contact the st | udy team to discuss |
| reviewed this research stud | on of Human Subjects at the l<br>ly. You may contact them for a<br>concerns, comments, or comp | any questions about your | rights as a research |
| | SIGNATURI | ES | |
| • • • | erstand the information given to udy. Your agreement to have borm to your child's school. | • | |
| Name of Child | | | |
| Name of Parent/<br>Guardian | Relationship to Child | Signature | Date |

Study Contact: Timothy Walker, PhD Telephone:

#UTHealth Houston IRB NUMBER: HSC-SPH-20-0861 IRB APPROVAL DATE: 07/31/2023